CLINICAL TRIAL: NCT02738736
Title: Clarifying Optimal Sodium Intake Project- Objective 1
Brief Title: Clarifying Optimal Sodium Intake Project
Acronym: COSIP-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University College Hospital Galway (Other)
Collaborators: European Research Council (Other); National University of Ireland, Galway, Ireland (Other)
Responsible Party: Principal Investigator, Dr Andrew Smyth, Dr., University College Hospital Galway
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRBCRFG-010416
Record Dates: First submitted 2016-04-04; First posted 2016-04-14 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Blood Pressure; Hypertension; Kidney Disease; Cardiovascular Disease
MeSH Terms: conditions — Hypertension; Kidney Diseases; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sodium Reduction (Experimental): In addition to usual care, those randomised to the intervention arm will receive specific counseling on behavioural and environmental factors that promote sodium reduction after randomization and at all post-randomisation visits, targeting sodium intake of <100mmol/day (<2.3g/day).
  Interventions: Behavioral: Sodium Reduction
- Usual Care (No Intervention): Participants randomized to usual care will also attend a dietitian-developed healthy eating guidance session but will not receive specific recommendations targeting sodium intake.

INTERVENTIONS:
Behavioral: Sodium Reduction — In addition to usual care, those randomised to the intervention arm will receive specific counseling on behavioural and environmental factors that promote sodium reduction after randomization and at all specified post-randomisation visits, targeting sodium intake of <100mmol/day (<2.3g/day). A research dietitian will develop the specific components of the intervention, based on standardised approaches to education interventions
  Arms: Sodium Reduction

SUMMARY:
Hypertension is a leading risk factor for cardiovascular disease (CVD) globally, accounting for 25-35% of the population-attributable fraction. Sodium (salt) intake is a key determinant of blood pressure, and reducing sodium intake has emerged as an important target for population-based interventions to prevent CVD. However, there is considerable uncertainty about the optimal level of sodium intake that is associated with lowest CV risk, and whether optimal levels differ for different populations and individuals. International and national guidelines recommend low sodium intake (<2.3g/day, or lower) in all persons, and advocate a population-wide approach to reducing sodium. Most of the world's population (~95%) consume between 3 and 6g/day of sodium (mean intake 4.0g/day), which means that most people will require a major change to their diet, to achieve the guideline target (<2g/day). While there is convincing evidence that high sodium intake (>5g/day) is associated with an increased risk of CVD, compared to low or moderate intake, the evidence that low sodium intake (<2.0g/day) is associated with a lower risk of CVD than moderate intake (2.0-5g/day) is inconsistent and inconclusive. The investigators plan to conduct a Phase IIb clinical trial to evaluate the role of low sodium intake (versus moderate) on cardiovascular biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 years or older
* Systolic blood pressure <160mmHg and diastolic blood pressure <95mmHg on three office blood pressure readings at time of screening and confirmed by a study ABPM before randomization of <150/90mmHg
* No change in anti-hypertensive or diuretic medications (including dose) for 3 months before screening visit
* Consumption of moderate sodium intake at screening, defined as an estimated daily sodium intake of >2.3/day estimated from food frequency questionnaire (FFQ)
* Self-reported willingness to modify dietary intake over sustained period, and adhere with directed recommendations over 2 years.
* Signed written informed consent

Exclusion Criteria:

* Known chronic kidney disease (CKD) or most recent eGFR ≤60ml/min/1.73m2
* Participants who are ineligible for COSIP based on their eGFR will be approached about entering the ongoing Sodium Intake in Chronic Kidney Disease (STICK) trial.
* Previous cardiovascular disease:

  * Myocardial infarction
  * Previous percutaneous coronary intervention (PCI) or percutaneous transluminal coronary angioplasty (PTCA)
  * Stroke (previous transient ischaemic attack [TIA] is not an exclusion criterion)
* Medical diagnosis known to be associated with abnormal renal sodium excretion, including the following:

  * Bartter syndrome
  * SIADH
  * Diabetes insipidus
* Serum sodium <125mmol
* Severe heart failure defined as NYHA Class III/IV OR left ventricular ejection fraction (LVEF) ≤30%
* High-dose loop or thiazide diuretic therapy, exceeding a total daily dose of frusemide 80mg, bumetanide 2mg, hydrochlorothiazide 50mg, bendroflumethiazide 2.5mg, indapamide 2.5mg, metolazone 2.5mg or the use of both a loop and thiazide diuretic
* Unable to follow educational advice of the research team
* Prescribed high-salt diet, low-salt diet or sodium bicarbonate
* Symptomatic postural hypotension or receiving treatment for postural hypotension
* Current or recent use (within one month) of immunosuppressive medications including tacrolimus, cyclosporine, azathioprine or mycophenolate mofetil
* Pregnancy or lactation
* Unable to comply with 24-hour urinary collections, or medical condition making collection of 24-hour urinary collection difficult (e.g. severe urinary incontinence)
* Participant unlikely to comply with study procedures or follow-up visits due to severe comorbid illness or other factor (e.g. inability to travel for follow-up visits, drug or alcohol misuse) in the opinion of the research team
* Cognitive impairment defined as a known diagnosis of dementia or inability to provide informed consent due to cognitive impairment in the opinion of the investigator
* Body Mass Index (BMI) <20 kg/m2 or BMI>40 kg/m2
* Participating in another clinical trial or previous allocation in this study

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2016-04; Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Change in cardiovascular biomarkers (Renin) | 24 months
  Change in renin from baseline to final follow-up, measured from serum measurements taken at randomisation and final visit (T8).
Change in cardiovascular biomarkers (Aldosterone) | 24 months
  Change in aldosterone from baseline to final follow-up, measured from serum measurements taken at randomisation and final visit (T8).
Change in cardiovascular biomarkers (Troponin T) | 24 months
  Change in troponin T from baseline to final follow-up, measured from serum measurements taken at randomisation and final visit (T8).
Change in cardiovascular biomarkers (Pro-BNP) | 24 months
  Change in Pro-BNP from baseline to final follow-up, measured from serum measurements taken at randomisation and final visit (T8).
Change in cardiovascular biomarkers ( C-reactive protein) | 24 months
  Change in C-reactive protein from baseline to final follow-up, measured from serum measurements taken at randomisation and final visit (T8).

SECONDARY OUTCOMES:
Change in 24-hour urinary sodium excretion | 24 months
  Change in 24-hour urinary sodium excretion from baseline to final visit (two years)
Change in mean systolic and diastolic blood pressure from 24-hour ambulatory blood pressure monitoring | 24 months
  Change in mean systolic and diastolic blood pressure from 24-hour ambulatory blood pressure monitoring completed at baseline and final visit (two years)
Change in functional status as measured by the assessment functional status questionnaire | 24 months
Change in eGFR (MDRD formula) | 24 months
  Change in eGFR (MDRD formula) from baseline to final follow-up
Change in eGFR(CKD-EPI formula) | 24 months
  Change in eGFR (CKD-EPI formula) from baseline to final follow-up
Change in RNA measured through PAXgene RNA blood samples | 24 months
Number of recorded falls, syncope and pre-syncope | 24 months
Number of cardiovascular events | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Martin J O'Donnell, MB PhD MRCPI, Principal Investigator — National University of Ireland, Galway; Andrew Smyth, MB PhD, Principal Investigator — National University of Ireland, Galway
Locations (1):
- HRB Clinical Research Facility Galway, Galway, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Smyth A, Judge C, Kerins C, McDermott S, Niland A, Corcoran C, Dineen R, Alvarez-Iglesias A, Nolan A, Mente A, Griffin MD, O'Shea P, Canavan M, Yusuf S, O'Donnell M. Dietary counselling to reduce moderate sodium intake: effects on cardiovascular and renal biomarkers: primary findings of the COSIP and STICK phase II feasibility randomised controlled trials. EClinicalMedicine. 2023 Feb 15;57:101856. doi: 10.1016/j.eclinm.2023.101856. eCollection 2023 Mar. PMID 37064508
- [Derived] Smyth A, Yusuf S, Kerins C, Corcoran C, Dineen R, Alvarez-Iglesias A, Ferguson J, McDermott S, Hernon O, Ranjan R, Nolan A, Griffin M, O'Shea P, Canavan M, O'Donnell M. Clarifying Optimal Sodium InTake In Cardiovasular and Kidney (COSTICK) Diseases: a study protocol for two randomised controlled trials. HRB Open Res. 2022 Feb 7;4:14. doi: 10.12688/hrbopenres.13210.2. eCollection 2021. PMID 36348660